CLINICAL TRIAL: NCT00946920
Title: An Open-Label, Multi-Centre, Randomised, Parallel-Arm One-Year Trial, Comparing the Efficacy and Safety of Degarelix Three-Month Dosing Regimen With Goserelin Acetate in Patients With Prostate Cancer Requiring Androgen Deprivation Therapy
Brief Title: A Trial of Degarelix in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FE200486 CS35; 2008-005276-27 (EudraCT Number)
Record Dates: First submitted 2009-07-03; First posted 2009-07-27 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Degarelix 240 mg/480 mg (Experimental)
  Interventions: Drug: Degarelix
- Goserelin acetate (Active Comparator)
  Interventions: Drug: Goserelin acetate

INTERVENTIONS:
Drug: Degarelix — The degarelix doses were administered by subcutaneous (s.c.) injections into the abdominal wall. A starting dose of 240 mg degarelix was administered on Day 0. One month later a maintenance dose of 480 mg was administered. This was repeated after 4, 7, and 10 months (ie a total of 5 administrations).
  Other Names: Firmagon; FE200486
  Arms: Degarelix 240 mg/480 mg
Drug: Goserelin acetate — The goserelin doses were administered by subcutaneous (s.c.) implants into the abdominal wall. An initial dose of 3.6 mg goserelin was administered on Day 0. One month later a subsequent dose of 10.8 mg was administered and this was repeated after 4, 7, and 10 months (ie a total of 5 implants).
  Other Names: Zoladex
  Arms: Goserelin acetate

SUMMARY:
A phase 3, open-label, parallel group, one year trial comparing the efficacy and safety of degarelix 3-month depot with the established therapy goserelin acetate 3-month implant in patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Has a histological confirmed prostate cancer Gleason graded).
* Has a screening testosterone above 2.2 ng/mL.
* Rising prostate-specific antigen (PSA).
* Has Eastern Cooperative Oncology Group (ECOG) score of ≤ 2.
* Has a life expectancy of at least one year.

Exclusion Criteria:

* Current or previous hormone therapy.
* Has received therapy with finasteride and dutasteride within 12 weeks and 25 weeks, respectively, prior to screening.
* Has a history of severe untreated asthma, anaphylactic reactions, or severe urticaria and/or angioedema.
* Has a heart insufficiency.
* Has a previous history or presence of another malignancy, other than prostate cancer or treated squamous/basal cell carcinoma of the skin, within the last five years.
* Has a clinically significant medical condition (other than prostate cancer) including, but not limited to, renal, haematological, gastrointestinal, endocrine, cardiac, neurological, or psychiatric disease and alcohol or drug abuse or any other condition which may affect the patient's health or the outcome of the trial as judged by the Investigator.
* Has received an investigational drug within the last 28 days before the Screening Visit or longer if considered to possibly influencing the outcome of the current trial.
* Is candidate for curative therapy, i.e. radical prostatectomy or radiotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (126):
- United States (36):
  - Urology Centers Of Alabama, Homewood, Alabama
  - Arkansas Urology, Little Rock, Arkansas
  - Urology Associates of Central CA, Fresno, California
  - Medresearch, La Mesa, California
  - South Orange County Medical Research Center, Laguna Hills, California
  - Atlantic Urology Medical Group, Long Beach, California
  - Anschutz Cancer Pavillion, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Urological Associates of Bridgeport, P.C., Trumbull, Connecticut
  - Urology Associates of Dover, PA, Dover, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - South Florida Medical Research, Aventura, Florida
  - Florida Foundation for Healthcare Research, Ocala, Florida
  - Georgis Patsias, MD, PA, Wellington, Florida
  - Palm Beach Urology Associates, PA, Wellington, Florida
  - Indiana University Department of Urology, Indianapolis, Indiana
  - Kansas City Urology Care, PA, Overland Park, Kansas
  - Urological Associates of Englewood, Englewood, New Jersey
  - Hamilton Urology PA, Hamilton, New Jersey
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Urology Group of New Mexico, PC, Albuquerque, New Mexico
  - Capital Region Urological Surgeons and Research Associates, Albany, New York
  - Hudson Valley Urology P.C., Poughkeepsie, New York
  - Metrolina Urology Clinic, Charlotte, North Carolina
  - Northeast Urology Research, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Alliance Urology Specialists, Greensboro, North Carolina
  - Urologic Consultants of SEPA, Bala-Cynwyd, Pennsylvania
  - State College Urologic Association, State College, Pennsylvania
  - Grand Strand Urology, Myrtle Beach, South Carolina
  - Urology Clinics of North Texas, PA, Dallas, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Urology of Virginia, Norfolk, Virginia
  - Virginia Urology Center, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - Seattle Urology Research Center, Burien, Washington
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Antwerpen, Edegem
  - UZ Gent, Ghent
  - AZ Groeninge - Campus Sint-Maarten, Kortrijk
- Canada (13):
  - Southern Interior Medical Research Inc., Kelowna, British Columbia
  - Dr. Cal Andreou Research, Surrey, British Columbia
  - Can-Med Clinical Research Inc., Victoria, British Columbia
  - Dr Gary Steinhoff Clinical Research, Victoria, British Columbia
  - Bramalea Medical Centre, Brampton, Ontario
  - Urology Associates / Urologic Medical Research, Kitchener, Ontario
  - Mor Urology, Inc., Newmarket, Ontario
  - Ivestigational site, Scarborough Village, Ontario
  - Anthony Skehan Medicine Professionals Corporation, Thunder Bay, Ontario
  - Bloor West Professional Center, Toronto, Ontario
  - The Health Institute for Men, Toronto, Ontario
  - Uro Laval, Laval, Quebec
  - Notre Dame Hopital, Montreal
- Czechia (8):
  - Urocentrum Brno, Brno
  - Nemocnice Jindrichuv Hradec, a.s., Jindřichův Hradec
  - Kromerizska nemocnice a.s., Kroměříž
  - Slezska nemocnice, Opava
  - Fakultni nemocnice v Motole, Praha 5, Prague
  - Fakultni Thomayerova nemocnice s poliklinikou, Praha 4, Prague
  - Vseobecna fakultni nemocnice v Praze, Praha 2, Prague
  - Krajska nemocnice T. Bati a.s., Zlín
- Finland (4):
  - Pietarsaaren sairaala/ Malmin terveydenhuoltoalue, Jakobstad
  - Pohjois-Karjalan keskussairaala, Joensuu
  - ODL Terveys Oy, Oulu
  - Tampereen yliopistollinen sairaala, Tampere
- Germany (4):
  - Investigational site, Aachen
  - Investigational site, Kirchheim
  - Klinikum Mannheim Universitätsklinikum GmbH, Mannheim
  - Urologische Studienpraxis, Nürtingen
- Hungary (9):
  - Fövárosi Önkormányzat Bajcsy-Zsilinszky Kórház, Budapest
  - Fövárosi Önkormányzat uzsoki utcai Kórház, Budapest
  - Semmelweis Egyetem, Budapest
  - Dombóvári Szent Lukács Egészségügyi Kht., Dombóvár
  - Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Miskolci Semmelweis Ignác Egészségügyi Központ és Egyetemi Oktató Kórház Nonprofit Kft, Miskolc
  - Pécsi Tudományegyetem, Pécs
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - Jávorszky Ödön Kórház, Vác
- Mexico (8):
  - Hospital Christus Muguerza del Parque, Chihuahua City, Chihuahua
  - Hospital Aranda de la Parra , S.A. de C.V., León, Guanajuato
  - Hospital Angeles Culiacan, Culiacán, Sinaloa
  - Consultorio de Especialidad en Urologia Privado, Durango, Durango
  - Centro Medico Dalinde, Mexico City
  - Hospital Angeles Lindavista, Mexico City
  - Operadora MSB, S.A. de C.V. (Medica Sur CIF-BIOTEC), Mexico City
  - Consultorio Medico, Zapopan, Jalisco
- Netherlands (4):
  - AMC, Amsterdam
  - Catharina-ziekenhuis, Eindhoven
  - Atrium MC, Heerlen
  - MC Haaglanden, The Hague
- Poland (5):
  - SPZOZ Wojewodzki Szpital Zespolony im. J.Sniadeckiego, Bialystok
  - Centrum Medyczne Medur Sp. z o.o., Bielsko-Biala
  - Gabinet Lekarski, Krakow
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku, Słupsk
  - LexMedica, Wroclaw
- Romania (10):
  - Private Medical Center, Arad
  - Brasov Emergency Clinical County Hospital, Brasov
  - "Fundeni" Clinical Institute, Bucharest
  - "Sfantul Ioan" Emergency Clinical Hospital, Bucharest
  - Dinu Uromedica, Bucharest
  - Prof. Dr. Th. Burghele Clinical Urology Hospital, Bucharest
  - PROVITA 2000 Medical Center, Constanța
  - "Dr. C.I. Parhon" Clinical Hospital, Lasi
  - Vita Care Flav Medical Center, Piteşti
  - Emergency County Clinical Hospital Sibiu, Sibiu
- Russia (9):
  - City Clinical Hospital #60, Moscow
  - Moscow State University of Medicine and Dentistry, Moscow
  - "Clinic Andros" LLC, Saint Petersburg
  - "Orkli" LLC, Saint Petersburg
  - City Hospital # 26, Saint Petersburg
  - City Hospital #15, Saint Petersburg
  - St. Petersburg State Medical University n.a. I.P. Pavlov, Saint Petersburg
  - St.Petersburg Multi-Field City Hospital #2, Saint Petersburg
  - Regional Clinical Oncology Center, Vladimir
- Ukraine (8):
  - Municipal Institution "Cherkasy Regional Oncology Dispensary", Cherkassy
  - Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Donetsk Regional Clinical Territorial Medical Association, Donetsk
  - Ivano-Frankivsk Regional Oncology Dispensary, Ivano-Frankivsk
  - Regional Clinical Center of Urology and Nephrology n.a. V.I.Shapoval, Kharkiv
  - Kyiv City Clinical Hospital #3, Kyiv
  - Odesa Regional Clinical Hospital, Odesa
  - Municipal Institution "Zaporizhzhia Regional Clinical Hospital", Zaporizhzhya
- United Kingdom (4):
  - Castle Hill Hospital, Cottingham
  - Ipswich Hospital, Ipswich
  - Royal Liverpool University Hospital, Liverpool
  - The Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met the eligibility criteria were randomized to degarelix or goserelin acetate treatment in a 2:1-ratio. 859 subjects were randomized but 11 subjects did not receive any treatment.
Period: Overall Study
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Started | 565 (Received at least one dose of degarelix.) | 283 (Received at least one dose of goserelin acetate.)
Full Analysis Set (FAS) | 565 (Received at least one dose of degarelix and had at least one post-dosing efficacy assessment.) | 282 (Received at least one dose of goserelin and had at least one post-dosing efficacy assessment.)
Completed | 455 | 239
Not Completed | 110 | 44
Not completed — Withdrawal by Subject | 28 | 15
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 5 | 2
Not completed — Adverse Event | 41 | 14
Not completed — Protocol Violation | 16 | 8
Not completed — Miscellaneous reasons | 18 | 3

BASELINE CHARACTERISTICS:
Population: FAS
Groups:
- Total: Total of all reporting groups
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate | Total
Number analyzed (Participants) | 565 | 282 | 847
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (8.3) | 71.1 (7.9) | 71.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 565 | 282 | 847
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 45 | 25 | 70
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 41 | 16 | 57
  White | 475 | 239 | 714
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Median Baseline Serum Testosterone Levels (ng/mL) [Median (Full Range); unit: ng/mL] | 4.52 [0.56 to 14.5] | 4.62 [0.07 to 13.2] | 4.54 [0.07 to 14.5]
Median Baseline Serum Prostate-specific Antigen Levels (ng/mL) [Median (Full Range); unit: ng/mL] | 19.0 [0.26 to 8762] | 19.1 [0.01 to 12961] | 19.0 [0.01 to 12961]
Baseline Short Form-36 (SF-36) Total Scores [Mean (Standard Deviation); unit: units on a scale] — The SF-36 is a multi-purpose, short-form health survey with only 36 questions and with a minimum score of 0 and a maximum score of 100. The higher score the better health. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. The SF-36 has proven useful in surveys of general and specific populations, comparing the relative burden of diseases, and in differentiating the health benefits produced by a wide range of different treatments.
  units on a scale | 49.7 (11.5) | 50.2 (11.4) | 49.9 (11.4)
Baseline Total International Prostate Symptom Scores (IPSS) [Mean (Standard Deviation); unit: units on a scale] — IPSS is used to assess severity of lower urinary tract symptoms and to monitor the progress of symptoms once treatment has been initiated. It contains 7 questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia. Each question is assigned a score of 0-5 (i.e. the minimum total score is 0 and the maximum is 35). A score of "0" corresponds to a response of "not at all" for the first six symptoms and "none" for nocturia, and a score of 5 corresponds to a response of "almost always" for the first six symptoms and "5 times or more" for nocturia.
  units on a scale | 11.8 (7.93) | 11.6 (8.02) | 11.7 (7.96)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Probability of Testosterone at Castrate Level (≤0.5 ng/mL) With Degarelix
Description: This co-primary outcome measure was used to demonstrate that degarelix is effective with respect to achieving and maintaining testosterone suppression to castrate levels, evaluated as the proportion of patients with testosterone suppression ≤0.5 ng/mL from Day 28 to Day 364.
Time Frame: From Day 28 to Day 364
Population: FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Degarelix 240 mg/480 mg
Number analyzed (Participants) | 565
percentage of participants | 90.0 [87.0 to 92.3]

2. Primary Outcome: Difference in Cumulative Probability of Testosterone at Castrate Level (≤0.5 ng/mL) Between Degarelix and Goserelin
Description: This co-primary outcome measure was used to establish non-inferiority of degarelix as compared to goserelin with regard to achieving and maintaining testosterone suppression at castrate levels (≤0.5 ng/mL) from Day 3 to Day 364, using a non-inferiority margin of 5 percentage points.
Time Frame: Day 3 to Day 364
Population: FAS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
percentage of participants | 85.0 [81.6 to 87.8] | 5.3 [3.1 to 8.4]
Statistical Analysis 1: Comparison: Degarelix 240 mg/480 mg vs Goserelin Acetate; The cumulative probability of testosterone ≤0.5 ng/mL from Day 3 to Day 364 was estimated by the Kaplan-Meier method. Only testosterone measurements taken at scheduled trial visits from Day 3 to Day 364 were included in the analysis. The hypothesis to test was the following: a non-inferiority assessment determined whether degarelix was non-inferior to goserelin with respect to the cumulative probability of testosterone ≤0.5 ng/mL from Day 3 to Day 364; Test type: Non-Inferiority or Equivalence — The non-inferiority limit for the difference between treatments (degarelix versus goserelin acetate) was chosen to be -5 percentage points; Kaplan-Meier estimate = 79.6, 95% CI 2-sided [75.6 to 83.7]

3. Secondary Outcome: Serum Levels of Testosterone Over Time
Description: Median testosterone levels are presented as absolute values at Baseline (in Baseline measures) and after 1, 2, 3, 6 and 13 months (below). One treatment month equals 28 days.
Time Frame: Baseline and after 1, 2, 3, 6 and 13 months
Population: FAS.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
ng/mL
  Month 1 | 0.10 [0.015 to 3.85] | 0.16 [0.04 to 1.77]
  Month 2 | 0.09 [0.015 to 0.41] | 0.10 [0.015 to 0.5]
  Month 3 | 0.09 [0.015 to 3.24] | 0.09 [0.015 to 5.4]
  Month 6 | 0.09 [0.015 to 1.57] | 0.09 [0.015 to 0.32]
  Month 13 | 0.11 [0.015 to 4.19] | 0.09 [0.015 to 0.95]

4. Secondary Outcome: Percent Change in Serum Levels of Prostate-specific Antigen (PSA) Over Time
Description: Serum PSA levels are presented as mean percent change from Baseline (in Baseline measures) after 1, 2, 3, 6 and 13 months. One treatment month equals 28 days.
Time Frame: Baseline and after 1, 2, 3, 6 and 13 months
Population: FAS.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
percent change
  Month 1 | -77 (23.7) | -57 (45.7)
  Month 2 | -89 (12.6) | -86 (18.1)
  Month 3 | -90 (15.4) | -86 (58.6)
  Month 6 | -90 (30.5) | -91 (18.2)
  Month 13 | -82 (104) | -77 (146)

5. Secondary Outcome: Change in Health-related Quality of Life (HRQoL), as Measured by Short Form-36 (SF-36) Score at Month 10 and Month 13 Compared to Baseline
Description: The SF-36 is a multi-purpose, short-form health survey with only 36 questions and with a minimum score of 0 and a maximum score of 100. The higher score the better health. It yields an 8-scale profile of functional health and well-being scores as well as psychometrically-based physical and mental health summary measures and a preference-based health utility index. The SF-36 has proven useful in surveys of general and specific populations, comparing the relative burden of diseases, and in differentiating the health benefits produced by a wide range of different treatments.
Time Frame: At baseline, 10 months and 13 months
Population: FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
units on a scale
  Month 10 | 0.52 (11.1) | 0.27 (10.6)
  Month 13 | 0.18 (10.9) | -0.87 (9.76)

6. Secondary Outcome: Change in International Prostate Symptom Score (IPSS) Score at Months 1, 4, 7, and 13 Compared to Baseline
Description: IPSS is used to assess severity of lower urinary tract symptoms and to monitor the progress of symptoms once treatment has been initiated. It contains 7 questions regarding incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia. Each question is assigned a score of 0-5 (i.e. the minimum total score is 0 and the maximum is 35). A score of "0" corresponds to a response of "not at all" for the first six symptoms and "none" for nocturia, and a score of 5 corresponds to a response of "almost always" for the first six symptoms and "5 times or more" for nocturia.
Time Frame: At baseline, 1 month, 4 months, 7 months and 13 months
Population: FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Number analyzed (Participants) | 565 | 282
units on a scale
  Month 1 | -1.06 (6.27) | -0.21 (6.22)
  Month 4 | -2.31 (6.65) | -1.74 (6.16)
  Month 7 | -2.47 (6.94) | -2.45 (6.80)
  Month 13 | -2.04 (7.28) | -1.52 (6.25)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from signed informed consent until the end-of-trial visit, Day 364 (Month 13).
Description: Adverse events were evaluated at each visit.
Arm/Group | Degarelix 240 mg/480 mg | Goserelin Acetate
Serious Adverse Events (participants affected / at risk) | 58/565 | 33/283
Other Adverse Events (participants affected / at risk) | 336/565 | 125/283
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Degarelix 240 mg/480 mg (N=565) | Goserelin Acetate (N=283)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 0
Cardiac failure acute (Cardiac disorders) | 2 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways (Infections and infestations) | 1 | 0
Injection site abscess (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Coronary artery reocclusion (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour local invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 3 | 1
Syncope (Nervous system disorders) | 3 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Degarelix 240 mg/480 mg (N=565) | Goserelin Acetate (N=283)
Hot flush (Vascular disorders) | 160 (175) | 76 (80)
Injection site pain (General disorders) | 173 (429) | 4 (4)
Injection site erythema (General disorders) | 122 (323) | 0 (0)
Injection site nodule (General disorders) | 51 (112) | 0 (0)
Weight increased (Investigations) | 26 (26) | 24 (24)
Urinary tract infection (Infections and infestations) | 24 (30) | 18 (24)
Fatigue (General disorders) | 26 (28) | 15 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (21) | 21 (27)
Hypertension (Vascular disorders) | 22 (24) | 18 (21)
Pyrexia (General disorders) | 31 (40) | 7 (7)
Injection site swelling (General disorders) | 34 (102) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.